CLINICAL TRIAL: NCT06771271
Title: A Multi-center, Non-Randomized, Open-label, Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7200220 in Monotherapy and in Combination With Ranibizumab Following Intravitreal Administration in Patients With Diabetic or Uveitic Macular Edema
Brief Title: A Study to Investigate RO7200220 as Monotherapy and in Combination With Ranibizumab in Participants With Diabetic and Uveitic Macular Edema
Acronym: DOVETAIL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP40899
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Macular Edema; Uveitic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: RO7200220 Monotherapy (Experimental): Participants with DME received multiple ascending doses of RO7200220 (two doses at the assigned dose level), as intravitreal (IVT) injection, every 6 weeks (Q6W) in multiple cohorts.
  Interventions: Drug: RO7200220
- Part 2: Expansion of RO7200220 Monotherapy (Experimental): Participants with DME who were anti-VEGF and corticosteroid IVT treatment-naive received three doses of RO7200220 monotherapy, as IVT injection, every 4 weeks (Q4W) in Part 2 cohorts.
  Interventions: Drug: RO7200220
- Part 3: RO7200220 in Combination with Ranibizumab (Experimental): Participants with DME received RO7200220 as IVT injection followed by ranibizumab, 0.5 milligrams (mg) as IVT injection in Part 3.
  Interventions: Drug: RO7200220; Drug: Ranibizumab
- Part 4: RO7200220 Monotherapy (Experimental): Participants with UME received multiple doses of RO7200220 (three doses at the assigned dose level), as IVT injection, Q4W in multiple cohorts.
  Interventions: Drug: RO7200220

INTERVENTIONS:
Drug: RO7200220 — RO7200220 was administered as IVT injection.
  Other Names: Vamikibart
Drug: Ranibizumab — Ranibizumab was administered as IVT injection.
  Arms: Part 3: RO7200220 in Combination with Ranibizumab

SUMMARY:
The purpose of this study was to assess the safety and tolerability of RO7200220 as monotherapy (diabetic macular edema [DME] or uveitic macular edema [UME] population) and in combination with ranibizumab (DME population only).

ELIGIBILITY:
Inclusion Criteria:

DME Participants:

* Diagnosis of Diabetes Mellitus (DM) (Type 1 or Type 2), as defined by the World Health Organization and/or American Diabetes Association
* Macular edema associated with DR defined as macular thickening by spectral domain optical coherence tomography (SD-OCT) involving the center of the macula: central subfield thickness (CST) of ≥325 μm with Spectralis.
* Decreased visual acuity (VA) attributable primarily to DME, with BCVA letter score of 73 to 19 letters (both inclusive) on Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts (20/40 -20/400 Snellen equivalent).
* Clear ocular media and adequate pupillary dilation to allow acquisition of good quality retinal images to confirm diagnosis.

UME Participants:

* Diagnosis of noninfectious uveitis (NIU) of any anatomical type (anterior, intermediate, posterior, panuveitis). Active and inactive NIU is allowed.
* Macular edema associated with NIU defined as macular thickening by SD-OCT involving the center of the macula: CST of ≥325 μm with Spectralis.
* Decreased VA attributable primarily to UME, with BCVA letter score of 78 to 19 letters (both inclusive) on ETDRS-like charts (20/32 - 20/400 Snellen equivalent).
* Sufficiently clear ocular media and adequate pupillary dilation to allow acquisition of good quality retinal images to confirm diagnosis.
* Either treatment naive or previously treated in the study eye or systematically (with washout periods and maximum doses applicable for specific treatments).

Exclusion Criteria:

* Any major illness or major surgical procedure within 1 month prior to Day 1
* Any febrile illness within 1 week prior to screening or Day 1
* Any stroke or myocardial infarction within 12 months prior to Day 1
* Any active proliferative DR (DME participants only)
* Panretinal photocoagulation or macular laser photocoagulation treatment prior to Day 1
* History of vitreoretinal surgery/pars plana vitrectomy
* Any cataract surgery within 3 months prior to Day 1 or any planned surgery during the study
* History of any glaucoma surgery including laser glaucoma procedures
* Uncontrolled glaucoma
* History of rubeosis iridis
* Any active ocular or periocular infection on Day 1
* Any presence of active intraocular inflammation on Day 1 or any history of intraocular inflammation (DME participants only)
* Any prior or concomitant periocular or IVT corticosteroids in the study eye (DME treatment naive participants only)
* Use of any systemic corticosteroids within 1 month prior to Day 1 (stable oral prednisone for UME participants allowed)
* Any prior or concomitant systemic anti-VEGF treatment within 6 months prior to Day 1
* Any concurrent use of biologics for immune-related diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Adverse Events (AEs) | Up to 18 weeks
Part 2: Number of Participants With Adverse Events (AEs) | Up to 24 weeks
Part 3: Number of Participants With Adverse Events (AEs) | Up to 20 weeks
Part 4: Number of Participants With Adverse Events (AEs) | Up to 36 weeks

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) | Part 1: Up to Week 18; Parts 2: Up to Week 24; Part 3: Up to Week 20; Part 4: Up to Week 36
Minimum Serum Concentration (Ctrough) | Part 1: Up to Week 18; Parts 2: Up to Week 24; Part 3: Up to Week 20; Part 4: Up to Week 36
Time to Peak Serum Concentration (Tmax) | Part 1: Up to Week 18; Parts 2: Up to Week 24; Part 3: Up to Week 20; Part 4: Up to Week 36
Area Under the Concentration-time Curve to the End of Dosing Period (AUC0-t) | Part 1: Up to Week 18; Parts 2: Up to Week 24; Part 3: Up to Week 20; Part 4: Up to Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (19):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - California Retina Consultants, Oxnard, California
  - Retina Institute of California Medical Group d/b/a Acuity Eye Group, Palm Desert, California
  - Byers Eye Insitute at Stanford, Palo Alto, California
  - Florida Eye Associates, Melbourne, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Illinois Retina Associates SC, Oak Park, Illinois
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - Sierra Eye Associates, Reno, Nevada
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon HSU, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Valley Retina Institute P.A., McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Univ of Virginia Ophthalmology, Charlottesville, Virginia
  - Karalis Johnson Retina Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No